CLINICAL TRIAL: NCT01757158
Title: Cesium-131 Seed Brachytherapy Plus Subtotal Resection for Lung Cancer Patients Who Are Not Candidates for Lobectomy or Patients With High Risk of Local Recurrence
Brief Title: Cesium-131 Seed Brachytherapy Plus Subtotal Resection for Lung Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: IsoRay Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0908010555
Record Dates: First submitted 2012-03-07; First posted 2012-12-28 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Lung Cancer
Keywords: lung cancer; lobectomy; local recurrence
MeSH Terms: conditions — Lung Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cs-131 brachytherapy seeds (Experimental): sub-lobar resection plus cesium-131 brachytherapy
  Interventions: Radiation: Cs-131 brachytherapy seeds

INTERVENTIONS:
Radiation: Cs-131 brachytherapy seeds — Cesium-131 is another radiation seed that may more effectively treat lung cancer patients. Cs-131 has been previously used in prostate cancer successfully. Cs-131 has similar energy to I-125 but has a much shorter half life (9days as compared to 60 days for I-125). Patients who receive Cs-131 radiation seeds are expected to be radioactive for 30 days (1 month) as compared to 180 days (6 months) with I-125.
  Other Names: Brachytherapy

SUMMARY:
The primary curative treatment of lung cancer patients is surgery, chemotherapy and/or radiation therapy (either or all depending on the extent of disease). Surgical resection usually requires removal of a lobe of the lung (lobectomy). There are, however, some patients who are unable to have a lobectomy. There are several reasons why a patient should not have a lobectomy including prior operations in the same area of the lung or poor lung functions. Sub-lobe operations (less than a full lobectomy), are alternatives for these patients. Types of sub-lobe operations include wedge resection or segmentectomy.

However, a randomized trial in early stage lung cancer patients that compared lobectomy versus wedge resection showed worse local control of cancer with wedge resection. Therefore, localized disease wedge resection is considered an inadequate operation. This inadequacy can be compensated if radiation seeds are added to the site of wedge resection. Iodine-125 (I-125) is the most commonly used radiation seed for this purpose. I-125, however, unfortunately has a relatively long half life (time taken for activity to become half) of 2 months. Therefore, the patient is technically 'radioactive' for an average of 6 months to 1 year. This can seriously compromise quality of life.

Cesium-131 is another radiation seed that may more effectively treat lung cancer patients. Cs-131 has been previously used in prostate cancer successfully. Cs-131 has similar energy to I-125 but has a much shorter half life (9days as compared to 60 days for I-125). Patients who receive Cs-131 radiation seeds are expected to be radioactive for 30 days (1 month) as compared to 180 days (6 months) with I-125. The objective of this study is the use Cs-131 radiation seeds in lung cancer patients who are planning to undergo a wedge resection for localized disease and follow the patients for cancer control and toxicity. These results will be compared to pre-existing data for I-125 treatment outcomes in lung cancer patients who have had a wedge resection for localized disease.

DETAILED DESCRIPTION:
A lobectomy (removal of a full lobe of the lung or removal of ¼ - 1/5 of the entire lungs) is a part of the primary curative treatment for people with lung cancer. There are, however, some patients who are unable to have a lobectomy. There are several reasons why a patient should not have a lobectomy including prior operations in the same area of the lung or poor lung functions. Sub-lobe operations (less than a full lobectomy), are alternatives for these patients. Types of sub-lobe operations include wedge resection or segmentectomy.

However, a randomized trial in early stage lung cancer patients that compared lobectomy versus wedge resection showed that cancer was not controlled as well in individuals who had the wedge resection. Localized disease wedge resection alone is therefore considered an inadequate operation. This inadequacy, however, can be compensated for if radiation seeds are implanted (added) to the site of wedge resection.

Iodine-125 radiation seeds are currently the most common radioactive material implanted in the operative bed after wedge resection. However, I-125 has a half-life of 60 days. This causes the patient to be "radioactive" for 6 months to 1 year. When an individual is radioactive they must take necessary precautions that result in a significantly compromised quality of life. These precautions are 1) no continuous close contact (less than 3 feet) for a significant duration of time (more than 15 minutes), 2) no close contact with pregnant women and children, 3) adequate precautions especially during air travel and 4) risk of radioactive seed displacement several months.

The local control of cancer with this treatment is >95%_ %. Cesium-131 is a novel radiation seed that has the same energy as I-125 but has a much shorter half life (9days). That means that Cs-131 seeds give off all their radiation at a faster rate. When a radioactive seeds gives off all of its radiation it is no longer radioactive and the dangers of radioactivity no longer exist. With a half life of 9 days, Cs-131 gives off all of its radiation in 1 month. This significantly reduces the time when the patient is 'radioactive'. Therefore, Cs-131 has less of a negative affect on quality of life than I-125.

In addition, because of Cs-131's significantly faster rate of radiation dissemination, faster growing cancers (especially lung cancer) cells should be killed more efficiently thereby increasing cancer control rates. In addition, the lesser total radiation time may result in reduced short term and long term side effects.

Cs-131 is FDA approved and has been used mostly for prostate cancer. Our experience with Cs-131 in prostate cancer has shown it to be a very well tolerated treatment with excellent cure rates.

The primary study endpoint is to assess local control of localized lung cancers after limited resection (wedge resection or segmentectomy) and Cs-131 seed placement in comparison to previously assessed local control of localized lung cancers after limited resection and I-125 seed placement. The primary objective is to assess local control after a wedge resection and Cs-131 implant. The secondary objective is to assess quality of life (as related to side effects) of Cs-131 seed placement after limited surgical resection in lung cancers and compare it to already existing data on I-125 tolerability.

Procedures that are part of regular cancer care and may be done whether a patient enrolls in the research study or not include:

1. CT scans of patient chest
2. Medistinoscopy (only if the surgeon is suspicious that there is cancer in the patient's lymph nodes),

   * If the cancer has spread to the lymph nodes, patients will no longer be eligible for the study as the classification of their disease would no longer be NSCLC. Patients would alternately receive appropriate, and standard treatment

Standard procedures being done only because the patient is part of the study;

1) Quality of life questionnaires

Follow-up Patients will be monitored for local recurrence, regional recurrence and distant recurrence and progression for three years.

Local recurrence: recurrence within the same lobe or hilum (N1 nodes), or at the staple line after treatment effects such as scarring have subsided.

Regional recurrence: recurrence within another lobe or pleura on the same side as the resection, or the ipsilateral mediastinal (N2) nodes.

Distant recurrence: recurrence within contralateral lobe, contralateral mediastinal (N3) nodes or distant metastatic disease (other organs).

Patients also will be monitored for additional primaries and regional recurrence, with histological confirmation whenever possible. Autopsy reports will be obtained whenever possible. A copy of the death certificate will also be obtained.

Protocol follow-up will be performed at 3, 6, 12, 18, 24, and 36 months and yearly to 5 years. The yearly follow-up visits for Years 4 and 5 will consist of either a phone call or clinical visit (at investigator's discretion) for vital status only. These follow-up visits will occur + 60 days from the yearly anniversary date of the resection.

A CT scan will be performed pre-operatively and at 3, 6, 12, 18, 24, 30 and 36 months.

QoL using the SF36 and UCSD Shortness of Breath Questionnaire will be obtained pre-operatively and at 3, 12 and 24 months.

Post-operative adjuvant chemotherapy may be given at the discretion of the treating physician. Postoperative adjuvant radiation therapy will never be performed.

Evaluation of Outcomes

Local Recurrence (primary endpoint)

Local recurrence is indicated when a follow-up examination shows growth of primary tumor or abnormality in the resected lobe on CT scan. Since scarring may occur adjacent to the brachytherapy site, a CT scan will be obtained at 3 months. This will form the baseline study that local recurrence will be judged against. Increased parenchymal opacification (by 25% or more) adjacent to the staple line/mesh line will be considered suspicious for local recurrence. The repeated CT scans should allow any significant changes to be observed even if there is a slight image artifact from the metal seeds which may interfere with interpretation of the CT scan.

Any suspicious areas will be confirmed by a needle biopsy.

Scans for Disease Relapse Unconfirmed by Biopsy If biopsy of suspicious areas is not feasible, then a PET scan is required. Copies of the PET scan, the 3- month (baseline) CT scan and the most current CT scan.

Quality of Life As a secondary outcome, patient-centered quality of life (QoL) data will be measured using the SF36 and dyspnea will be measured using the UCSD Shortness of Breath Questionnaire. [Eakin, 1998] These are ill patients with significant pulmonary morbidity. It will be important to quantify any changes in overall health and pulmonary-specific symptoms in this population. Each patient will act as his or her own control. These validated instruments have been used in many trials of patients with severe lung disease. Measurements will be undertaken before and at 3, 12 and 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have suspicious lung nodule for clinical stage I/recurrent Lung Cancer
2. Mass Tumor size < 7 cm
3. Patient must have a CT scan of the chest with upper abdomen within 90 days prior to date of pre-registration.
4. Patient must have ECOG/Zubrod performance status 0,1, or 2.
5. Resected lung cancers with positive margins

Exclusion Criteria:

1. Patient has already received high dose radiation to the area
2. Cancerous nodule is very close to the esophagus or spinal chord, thereby increasing the risk of radiation treatment
3. Pregnancy or unwillingness to practice a form of birth control (i.e. abstinence, oral contraceptives, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 5 years
  To assess local recurrence rate after a wedge resection and Cs-131 implant.

SECONDARY OUTCOMES:
Quality of Life | pre-surgery, 3 months, 12 months, 24 months
  To assess quality of life (as related to side effects) of Cs-131 seed placement after limited surgical resection in lung cancers and compare it to already existing data on I-125 tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Bhupesh Parashar, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any individual participant data for this trial as it has not accrued any patients and is now closed.